CLINICAL TRIAL: NCT06765395
Title: Applying Machine Learning to Explore Association Models Between Environmental Hormones, Breast Cancer, and a Dietary and Health Education Improvement Program: An Investigative Study
Brief Title: Explore Association Models Between Environmental Hormones andBreast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Pei-Hung Liao (Other)
Responsible Party: Sponsor-Investigator, Pei-Hung Liao, Associate professor, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Other Study IDs: (956)111-35
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Breast Diseases; Breast Adenocarcinoma
Keywords: Machine learning; association model; environmental hormones; breast cancer
MeSH Terms: conditions — Breast Diseases; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
investigated the association model between environmental hormone-related living habits and breast cancer, as well as dietary improvement programs through machine learning and clinical validation of patients with breast cancer.

DETAILED DESCRIPTION:
Female breast cancer is the second most common cancer worldwide and the age at diagnosis is decreasing. Traditional risk factor screening for breast cancer focuses on reproductive history, family history, age at menarche, and age at menopause; however, young patients diagnosed with breast cancer who do not meet the above risk factors are becoming common.This study established an association model between environmental hormones and breast cancer through machine learning to improve dietary programs to reduce the incidence of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients aged 20 years or above; (2) patients with breast cancer.

Exclusion Criteria:

* non-patients with breast cancer

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study recruited research subjects from an outpatient clinic and ward of the Department of General Surgery of the Cheng Hsing General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 687 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
established an association model between environmental hormones and breast cancer | 2015~2024
  The basic personal information of the participants included gender, age, height, weight, past disease history, family history, reproductive history, postoperative medication, chemotherapy type, breast cancer pathology type, stage, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei university of Nursing and health science, Taipei, Peitou, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang CY, Su CH, Chang CH, Ho CS, Liao PH. Applying machine learning to explore association models between environmental hormones, breast cancer, and a dietary and health education improvement program: an investigative study. Int J Environ Health Res. 2025 Oct 16:1-10. doi: 10.1080/09603123.2025.2576144. Online ahead of print. PMID 41103105